CLINICAL TRIAL: NCT00964002
Title: A Phase II Trial to Assess the Efficacy of Efavirenz in Metastatic Patients With Androgen-independent Prostate Cancer
Brief Title: Efavirenz in Treating Patients With Metastatic Prostate Cancer
Acronym: FAVE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Bergonié (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000641767; IB-FAVE; IB 2008-23; INCA-RECF0889; EUDRACT-2008-002730-30
Record Dates: First submitted 2009-08-21; First posted 2009-08-24 (Estimated); Results first posted 2022-05-16 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2021-11

CONDITIONS: Prostate Cancer
Keywords: recurrent prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — efavirenz

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Efavirenz (Experimental): Patients will receive efavirenz 600 mg daily as oral tablets at bedtime and in fast condition (1-2 hours far from dinner) until objective biological, radiological or clinical disease progression or study discontinuation (withdrawal of consent or when the patient meets one criterion for treatment discontinuation).
  Individual dose escalation will be possible: if biological progression occurs at month 3, dose could be increased to 1200 mg/day in asymptomatic and non radiological progression patients (by step of 200 mg every 15 days).
  Interventions: Drug: efavirenz

INTERVENTIONS:
Drug: efavirenz

SUMMARY:
RATIONALE: Efavirenz may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase II trial is studying how well efavirenz works in treating patients with metastatic prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the effect of efavirenz on the PSA non-progression rate at 3 months in patients with castration-refractory metastatic prostate cancer.

Secondary

* To assess the effect of efavirenz on the PSA non-progression rate at 6 months.
* To assess the effect of efavirenz on overall survival.
* To assess the effect of efavirenz on PSA progression-free survival..
* To assess the tolerability and safety profile of efavirenz.

OUTLINE: This is a multicenter study.

Patients receive oral efavirenz once daily in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed prostate cancer

  * Metastatic disease
  * Castration-refractory disease
* No clinical symptoms related to disease progression

PATIENT CHARACTERISTICS:

* WHO performance status 0-2

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2008-05 (Actual); Primary Completion 2011-09-19 (Actual); Study Completion 2014-04-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nadine Houede, Principal Investigator — Institut Bergonié
Locations (1):
- Institut Bergonie, Bordeaux, France

REFERENCES:
- [Result] Houede N, Pulido M, Mourey L, Joly F, Ferrero JM, Bellera C, Priou F, Lalet C, Laroche-Clary A, Raffin MC, Ichas F, Puech A, Piazza PV. A phase II trial evaluating the efficacy and safety of efavirenz in metastatic castration-resistant prostate cancer. Oncologist. 2014 Dec;19(12):1227-8. doi: 10.1634/theoncologist.2014-0345. Epub 2014 Oct 29. PMID 25355844

RESULTS

PARTICIPANT FLOW:
Groups:
- Efavirenz: Patients will receive efavirenz 600 mg daily as oral tablets at bedtime and in fast condition (1-2 hours far from dinner) until objective biological, radiological or clinical disease progression or study discontinuation (withdrawal of consent or when the patient meets one criterion for treatment discontinuation).
  Individual dose escalation will be possible: if biological progression occurs at month 3, dose could be increased to 1200 mg/day in asymptomatic and non radiological progression patients (by step of 200 mg every 15 days). As dose increase is protocol/standard and we are not in a dose escalation trial (Phase I), patients with dose escalation will not be described or analyzed for the primary endpoint.
Period: Overall Study
Arm/Group | Efavirenz
Started | 61
Assessable for Safety | 59 (59 patients were assessable for safety, they received treatment at least once.)
Completed | 53
Not Completed | 8
Not completed — Protocol Violation | 8

BASELINE CHARACTERISTICS:
Groups:
- Efavirenz: Patients will receive efavirenz 600 mg daily as oral tablets at bedtime and in fast condition (1-2 hours far from dinner) until objective biological, radiological or clinical disease progression or study discontinuation (withdrawal of consent or when the patient meets one criterion for treatment discontinuation).
  Individual dose escalation will be possible: if biological progression occurs at month 3, dose could be increased to 1200 mg/day in asymptomatic and non radiological progression patients (by step of 200 mg every 15 days).
  efavirenz
Arm/Group | Efavirenz
Number analyzed (Participants) | 61
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 71 [67 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 61
Region of Enrollment [Count of Participants; unit: Participants]
  France | 61

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Without Prostate-specific Antigen Progression at 3 Months
Description: Prostate-specific antigen (PSA) non-progression rate is defined as the rate of patients with the absence of PSA progression.
  PSA progression is defined as follows :
  * In patients whose PSA has not decreased, progressive disease is a 25% increase over the baseline (on-study) and an increase in the absolute-value PSA level by at least 5 ng/mL, which is confirmed by a second value.
  * In patients whose PSA has decreased but has not reached response criteria, progressive disease would be considered to have occurred when PSA increases 25% over the nadir, provided that the increase is a minimum of 5 ng/mL and is confirmed.
  For the 3-month evaluation, patients who died within the 3 first months will be considered as progressions.
  PSA assessment is to be performed every 28 days in the first 6 months after inclusion then every 3 months until progression or end of treatment. PSA assessment to establish eligibility is to be obtained from the same local laboratory using the same PSA assay.
Time Frame: 3 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Efavirenz
Number analyzed (Participants) | 53
percentage of participants | 28.3 [16.8 to 42.3]

2. Secondary Outcome: Percentage of Participants Without Prostate-specific Antigen Progression at 6 Months
Description: Prostate-specific antigen (PSA) non-progression rate is defined as the rate of patients with the absence of PSA progression.
  PSA progression is defined as follows :
  * In patients whose PSA has not decreased, progressive disease is a 25% increase over the baseline (on-study) and an increase in the absolute-value PSA level by at least 5 ng/mL, which is confirmed by a second value.
  * In patients whose PSA has decreased but has not reached response criteria, progressive disease would be considered to have occurred when PSA increases 25% over the nadir, provided that the increase is a minimum of 5 ng/mL and is confirmed.
  For the 6-month evaluation, patients who died within the 6 first months will be considered as progressions.
  PSA assessment is to be performed every 28 days in the first 6 months after inclusion then every 3 months until progression or end of treatment. PSA assessment to establish eligibility is to be obtained from the same local laboratory using the same PSA assay.
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Efavirenz
Number analyzed (Participants) | 53
percentage of participants | 11.3 [4.3 to 23]

ADVERSE EVENTS:
Description: Only serious adverse events were monitored. Adverse events (non-serious) were not assessed/monitored during the study.
Arm/Group | Efavirenz
Serious Adverse Events (participants affected / at risk) | 11/59
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Efavirenz (N=59)
Psychosis (Psychiatric disorders) | 2 (2)
Confusion (Psychiatric disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Aortic injury (Injury, poisoning and procedural complications) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes